CLINICAL TRIAL: NCT00163865
Title: A Pilot Study of Boredom in a Community Sample of Adolescents and a Clinical Sample of Adolescents
Status: Completed | Type: Observational
Sponsor: Bayside Health (Other Government)
Collaborators: The Alfred (Other)
Responsible Party: Sponsor
Other Study IDs: BA 46/05
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2005-09

CONDITIONS: Mental Disorders; Affective Disorders; Anxiety Disorders; Attention Deficit and Disruptive Behavior Disorders; Psychotic Disorders
Keywords: Boredom; Adolescent; Mental illness; Depression; Anxiety
MeSH Terms: conditions — Mental Disorders; Mood Disorders; Anxiety Disorders; Attention Deficit and Disruptive Behavior Disorders; Psychotic Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Clinical Group: clinical adolescent group
- Community Group: community adolescent group

SUMMARY:
The aim of the following pilot study is to examine boredom in a community sample of adolescents and a clinical sample of adolescents. This is important in order to examine differences among healthy adolescents and adolescents with mental illness.

DETAILED DESCRIPTION:
Boredom has been recognized as a significant problem in a wide variety of areas. However, limited research has been focused on this construct (Vodanovich & Watt, 1999). Research into boredom in adolescents is especially lacking in the psychological literature. This is surprising given that adolescence is a time marked by change, stress, and identity issues.

The aim of the following pilot study is to examine boredom in a community sample of adolescents and a clinical sample of adolescents. This is important in order to examine differences among healthy adolescents and adolescents with mental illness, such as depression, anxiety, and ADHD. This has implications for both prevention and intervention strategies and programs, such as the assessment and treatment of adolescents with mental illness. Hence, the results of this study will be important in providing an evidence-based practice in the treatment of mental illness in adolescents.

Participants will be asked to complete one survey, the Boredom Proneness Scale (Farmer & Sundberg, 1986), and a demographic background form to measure gender, date of birth, country of birth, etc. The community sample of adolescents will be recruited from secondary schools in Victoria. The clinical sample of adolescents will be recruited from the Alfred Child and Adolescent Mental Health Service. It is envisaged that about 100 adolescents from each sample will be recruited to participate.

ELIGIBILITY:
Inclusion Criteria:

* 13-18 years of age
* has consenting guardian

Exclusion Criteria:

* unable to sufficiently understand self report measure
* IQ < 70

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2005-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Boredom proneness scale | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Campbell R Thorpe, MBBS FRANZCP, Principal Investigator — Alfred Hospital Bayside Health
Locations (1):
- Alfred Child and Adolescent Mental Health Service, Melbourne, Victoria, Australia